CLINICAL TRIAL: NCT03870724
Title: Women and Risk of Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Norwegian Diabetes Association (Other)
Responsible Party: Principal Investigator, Christin Waage, Postdoctor, University of Oslo
Other Study IDs: 2018/2517
Record Dates: First submitted 2019-02-27; First posted 2019-03-12 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Prevention; Cardiovascular diseases; Physical activity; Ethnic differences in health; Risk factors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a follow-up survey of women, 10-12 years after they were included in the population-based Stork Groruddalen study of pregnant women, primarily set up to study gestational diabetes and related health issues in pregnancy in a multiethnic population. The investigators will now update the information about the health status of these women to study the development of risk factors for type 2 diabetes and cardiovascular diseases.

DETAILED DESCRIPTION:
The STORK-Groruddalen is a cohort study of 823 pregnant women. Participation rate was high due to facilitation for ethnic minorities and data collection at the local Health Centres, set up to study ethnic differences in health to inform prevention strategies to reduce these differences. The investigators have published many papers from this well charatertized cohort, about gestational diabetes and related health issues in pregnancy. Participants have agreed to be contacted for subsequent follow-up surveys.

The inivestigators are now planning a follow-up study of these woman during 2019-2022, to study trajectories for risk factors for type 2 diabetes and cardiovascular diseases such as BMI, blood pressure, lipids, behavioural factors, physical activity and mental health and other health issues. The investigators will collect selfreported information through questionnaires, perform clinical measurements and take blood samples and buccal swabs. Collecting updated information about a range of health outcomes for women in this cohort will, together with already collected data, enable us to study the development of risk factors for type 2 diabetes and cardiovascular diseases in a life course perspective.

ELIGIBILITY:
Inclusion Criteria:

* Previous participants in the STORK G study still living in Norway

Exclusion Criteria:

* Moved out of Norway

Ages: 27 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Middle aged women, previous participants in the STORK G study still living in Norway
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes | 2 years
  Prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Anne Karen Jenum, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Faculty of Medicine, Institute of Health and Society, Oslo, Norway

REFERENCES:
- [Derived] Waage CW, Jenum AK, Mdala I, Lee-Odegard S, Braend AM, Sletner L, Berg JP, Birkeland KI. Diabetes and prediabetes among women universally screened for gestational diabetes: a multi-ethnic, population-based, prospective study with eleven years follow-up. BMC Public Health. 2025 Apr 3;25(1):1264. doi: 10.1186/s12889-025-22493-x. PMID 40181282
- [Derived] Waage CW, Toftemo I, Braend AM, Sletner L, Sommer C, Birkeland KI, Richardsen KR, Shakeel N, Vollestad NK, Jenum AK. Cohort profile update: the Norwegian STORK Groruddalen (STORK G) pregnancy and birth cohort-the role of ethnicity and causal pathways for obesity, type 2 diabetes, cardiovascular disease and other health issues. BMJ Open. 2023 Oct 29;13(10):e076251. doi: 10.1136/bmjopen-2023-076251. PMID 37899145